CLINICAL TRIAL: NCT04758156
Title: Comparison Between a 1L of Polyethylene Glycol+Ascorbic Acid as a Split Dose Bowel Preparation for Colonoscopy: Prospective, Randomized, Parallel, Multi-center Trial
Brief Title: Comparison Between a 1L of Polyethylene Glycol+Ascorbic Acid as a Split Dose Bowel Preparation for Colonoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jung Lee, Assistant Professor, MD, PhD, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1905-1831
Record Dates: First submitted 2021-02-15; First posted 2021-02-17 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Colon Adenoma; Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CleanViewAL (Experimental): 1L polyethylene glycol+ascorbic acid split dose
  Interventions: Drug: CleanViewAL
- SUPREP (Placebo Comparator): Oral sulfate solutiom
  Interventions: Drug: SUPREP

INTERVENTIONS:
Drug: CleanViewAL — 1L PEG + ascorbic acid bowel preparation for colonoscopy
  Arms: CleanViewAL
Drug: SUPREP — Oral sulfate solution for colonoscopy bowel preparation
  Arms: SUPREP

SUMMARY:
Comparison between a 1L of polyethylene glycol+ascorbic acid as a split dose and oral sulfate solution bowel preparation for colonoscopy

study design: prospective, randomized, parallel, multi-center trial in 3 hospitals in Korea ( Seoul National University hospital, Seoul National University Bundang hospital, Seoul Metropolitan Government-Seoul National University )

patient inclusion criteria

- aged 20-75 adults (out-clinic patients) scheduled for colonoscopy for any indication within the normal process of care

ELIGIBILITY:
Inclusion Criteria:

* Adult out clinic patients scheduled for colonoscopy for any indication within the normal process of care

Exclusion Criteria:

* previous history of significant gastrointestinal surgeries (except for appendectomy)
* known or clinically suspicious Inflammatory bowel disease patients
* known or suspected ileus/ GI obstruction
* previous history of major cancer or currently on treating cancer
* Major cardiovascular disease, respiratory disease, liver, hematologic diseases with complication
* severe cognitive impairment / dementia / confusion state
* past history within the last 12 months or current episode of severe constipation severe constipation
* Regular use of laxatives or colon motility-altering drugs (i. e. more than 2 - 3 times per week) in the last 28 days prior to screening and/or laxative use within 72 hours prior to administration of the preparation)
* women who are pregnant or lactating
* known phenylketonuria, glucose-6-phosphate dehydrogenase deficiency
* those who were allergic to any preparation components.
* those who, in the opinion of the investigator, should not be included in the study for any reason

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (BBPS) | at the time of colonoscopy procedure
  Bowel cleansing score

SECONDARY OUTCOMES:
questionnaire gathered for Tolerability, compliance, satisfaction | on the 1 day of colonoscopy via questionnaire
  information gathered via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jong Pil Im, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No